CLINICAL TRIAL: NCT01892618
Title: A Randomized Phase III Trial to Determine Whether Conjugated Pneumococcal Vaccine Can Improve the Immune Responsiveness Compared to Polyclonal Pneumococcal Vaccine in Patients With Untreated Chronic Lymphocytic Leukemia
Brief Title: Pneumococcal Vaccine in Untreated CLL Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Kimby, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-012642-22
Record Dates: First submitted 2013-06-12; First posted 2013-07-04 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — 13-valent pneumococcal vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pneumovax (Active Comparator): Pneumovax, 1x 0.5 ml injection
  Interventions: Drug: Pneumovax
- Prevenar 13 (Experimental): Prevenar 13, 1x 0.5 ml injection
  Interventions: Drug: Prevenar 13

INTERVENTIONS:
Drug: Prevenar 13 — 13-valent pneumococcal conjugated vaccine
  Arms: Prevenar 13
Drug: Pneumovax — 23-valent pneumococcal polysaccharide vaccine
  Arms: Pneumovax

SUMMARY:
The purpose of the study is to determine whether patients with chronic lymphocytic leukaemia (CLL) will benefit from vaccination with a 13-valent conjugated pneumococcal vaccine, Prevenar13, compared with a conventional 23-valent capsular polysaccharide vaccine in terms of immune response.

ELIGIBILITY:
Inclusion Criteria:

* Untreated CLL patients all Rai stages (0 to IV), as early as possible after diagnosis, always before any therapy with monoclonal antibodies and/or chemotherapy

Exclusion Criteria:

* Immunosuppressive therapy planned to start within 1 month
* Other malignancies
* Corticosteroids or other immunosuppressive drugs
* Previous allergic reaction to any vaccination in the past
* Neutropenia (PMNs < 500 cells/mm3)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Immune response to Pneumovax compared to immune response to Prevenar | 1 month post vaccination

SECONDARY OUTCOMES:
Serotype-specific immunoglobulin G (IgG) antibody levels | 1 and 6 months post vaccination
  Immune response to Pneumovax vs. Prevenar13
Levels of opsonophagocytic antibodies (OPA) | 6 months post vaccination
  Immune response
Serotype-specific IgG antibody levels by ELISA, geometric mean concentrations (GMCs)between arms | 1 and 6 months post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Eva Kimby, Professor, Principal Investigator — Karolinska University Hospital, SE-141 86 Stockholm, Sweden
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Zorger AM, Hirsch C, Baumann M, Feldmann M, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with haematological malignancies. Cochrane Database Syst Rev. 2025 May 21;5(5):CD015530. doi: 10.1002/14651858.CD015530.pub2. PMID 40396505